CLINICAL TRIAL: NCT03653897
Title: Performance of the ID-Cap System, in the Clinical Setting as an Aid to Measure Medication Adherence (DO Trial 2.0)
Brief Title: Performance of the ID-Cap System, an Ingestion Event Marker, in the Clinical Setting as an Aid to Measure Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EtectRX, Inc. (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ERX002
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
Keywords: Ingestion event marker; Ingestible sensor; Medication adherence; ID-Cap Medication Adherence Feedback System
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: This study is a prospective, open label, clinical study evaluating the safety and effectiveness of the ID-Cap System under direct observation in the clinical setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ID-Capsules- Active (Experimental): Subjects will ingest ID-Capsules containing the ingestible sensor which emits a signal from within the subject's stomach. This signal is detected by the wearable Reader, and the ingestion event is recorded.
  Interventions: Device: ID-Capsule- Active; Device: Wearable Sensor

INTERVENTIONS:
Device: ID-Capsule- Active — A standard gelatin or HPMC capsule with an embedded ingestible wireless sensor.
Device: Wearable Sensor — Subjects will wear an ID-Reader

SUMMARY:
The ID-Cap System is classified as an ingestion event marker (IEM), a Class II medical device. The system is intended to record time-stamped ingestions with the ingestible sensor, ID-Tag which transmits a signal to a wearable device, the ID-Cap Reader. In this study, 12-18 subjects will ingest capsules containing ingestible sensors while wearing the Reader and being observed in a clinic setting.

ELIGIBILITY:
Enrollment will be stratified to include at least two study participants in each BMI-Gender category. The BMI-Gender categories will be: Normal/Underweight (BMI<25), Overweight (BMI 25.0 to <30), and Obese (BMI>30.0); and Male/Female.

Inclusion Criteria:

* Men and women 18 years of age or older.
* For females of childbearing potential, negative urine pregnancy test at time of entry and assurance that a medically-accepted means of contraception will be used for the duration of the study.
* Able and willing to provide informed consent.
* Willing to adhere to all protocol requirements and study procedures.
* Adequate organ function at screening.

Exclusion Criteria:

* Unable to take oral medications.
* Women who are pregnant, breast-feeding, or plan to become pregnant during the study, and females of childbearing potential who are not using a medically-accepted means of contraception.
* Medical condition which may affect passage through the gastrointestinal tract (including, but not limited to, small bowel tumors, symptomatic intestinal adhesions, symptomatic active ulcerations, and radiation enteritis).
* Known hypersensitivity to any component of the ingestible ID-Capsule (including, but not limited to, gelatin, polyimide, magnesium, or silver).
* Significant medical condition, psychiatric condition, current alcohol or drug abuse, or other condition which may preclude the study participant from being able to follow study procedures or to safely participate in the opinion of the investigator.
* Participation in an investigational product study (e.g., medical device or drug study) within 30 days prior to screening, or prior participation in an Ingestion Event Marker study.
* Presence of an active implantable electronic medical device.
* Positive screen for drugs of abuse (detection of drug for which a valid prescription exists is not exclusionary).
* Any laboratory test result deemed clinical significant by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender at birth
Enrollment: 13 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Positive Detection Accuracy (PDA) | Up to 6 days
  The number of active ingestible sensors detected divided by the number of active ingestible sensors administered under direct observation.
Negative Detection Accuracy (NDA) | Up to 6 days
  The number of inactive empty capsules not detected divided by the number of inactive empty capsules administered under direct observation. Determination of NDA will also include the number of monitoring periods with no ingestion events detected by the Reader divided by the number of specific monitoring periods performed for the purpose of detecting false positives.

SECONDARY OUTCOMES:
Number of Study Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 6 days during ingestion events through the follow-up assessment scheduled within 3 to 5 days of the last ingestion]
  Incidence of mild, moderate, and severe adverse events overall and related to the device; discontinuations due to adverse events

OTHER OUTCOMES:
Detection Time | Up to 60 minutes post ingestion
  Time from ingestion of ID-Capsule to first detection by the ID-Cap Reader
Signal Duration | Up to 60 minutes post ingestion
  Time from first to last detection of the signal from the ingested sensor by the ID-Cap Reader

CONTACTS AND LOCATIONS:
Overall Officials: Gary Connor, RN, Study Director — EtectRX, Inc.
Locations (1):
- Quotient Sciences, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No